CLINICAL TRIAL: NCT04412512
Title: VATS Versus Thoracotomy for Pulmonary Hydatid Disease
Acronym: VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hassan II University (Other)
Responsible Party: Principal Investigator, Sara WAGUAF, Principal Investigator, Hassan II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VATS for pulmonary hydatid
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Hydatid Cyst
Keywords: pulmonary hydatid cyst; video-assisted thoracic surgery; thoracotomy
MeSH Terms: conditions — Echinococcosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: study the effect of a treatment and evaluate outcome postoperative
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VATS approach (Experimental): patients treated by VATS technique.
  Interventions: Procedure: VATS approach
- Thoracotomy approach (Active Comparator): patients treated by Thoracotomy technique
  Interventions: Procedure: Thoracotomy approach

INTERVENTIONS:
Procedure: VATS approach — video-assisted thoracic surgery approach
  Arms: VATS approach
Procedure: Thoracotomy approach
  Arms: Thoracotomy approach

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of minimally invasive surgery and compare the outcomes with patients undergoing thoracotomy in treatment of Pulmonary Hydatid Cyst.

Disease : pulmonary hydatid cyst.

Intervention:

* Group 1 : VATS approach.
* Group 2 : thoracotomy approach.

DETAILED DESCRIPTION:
After being informed about the study and the approach, all patients giving written informed consent to determine eligibility for study entry.

ELIGIBILITY:
Inclusion Criteria:

- all patients underwent surgery for pulmonary hydatid cyst

Exclusion Criteria:

* none

Ages: 6 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  evaluate the complication at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: sara WAGUAF, Principal Investigator — Hassan II University
Locations (1):
- Hassan II University, Casablanca, Morocco